CLINICAL TRIAL: NCT01227330
Title: Pilot Program to Improve Statin Adherence and Lower Cholesterol in Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU HSIRB 1174637
Record Dates: First submitted 2010-10-13; First posted 2010-10-25 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Hypercholesterolemia; Medication Adherence
MeSH Terms: conditions — Hypercholesterolemia; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medication adherence intervention (Experimental): Receives 12-week behavioral feedback intervention to improve adherence to statin medication
  Interventions: Behavioral: Medication adherence intervention
- Control (No Intervention): No intervention
- Attention-control (Active Comparator): Receives visits on the same schedule as the intervention group, with health education that is unrelated to medications or cholesterol
  Interventions: Behavioral: Attention-control

INTERVENTIONS:
Behavioral: Medication adherence intervention — 12-week behavioral feedback intervention to improve adherence to statin medication
  Arms: Medication adherence intervention
Behavioral: Attention-control — Health education visits that are unrelated to medications or cholesterol, provided on the same visit schedule as the intervention group
  Arms: Attention-control

SUMMARY:
The purpose of this study is to pilot test a behavioral medication adherence (MA) intervention compared to control condition in older adults with low adherence to medication for hypercholesterolemia.

DETAILED DESCRIPTION:
This study will answer the following primary research question:

1. What is the estimated effect size of a behavioral MA intervention on MA rates in older adults who are poorly adherent to statin medications?

   The study will also explore the following secondary research questions:
2. What is the estimated effect size of a behavioral MA intervention on low-density lipoprotein cholesterol (LDL-C) levels in older adults?
3. What is the estimated effect size of a behavioral MA intervention on high-density lipoprotein cholesterol (HDL-C) levels in older adults?
4. What is the feasibility of successfully testing this intervention protocol in a population of older adults with low adherence to statin medications?

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older at the time of study entry,
* Take a once-daily prescription statin medication for ≥ 6 months with no changes to statin prescription for at least 30 days prior to study entry,
* A score of ≤ 9 on the Short Blessed Test,
* Participants must self-administer his or her own medications without prompts from any other person or device.
* Baseline medication adherence rate of ≤ 90%.
* Participants agree to complete all study contacts and measurements, including the use of a special medication bottle with a Medication Event Monitoring System (MEMS) cap for the duration of the study.
* Able to open and close MEMS caps.

Exclusion Criteria:

* Participant's medications are managed by someone other than the participant
* Participant is unable or unwilling to use MEMS caps.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 6 months

SECONDARY OUTCOMES:
Serum cholesterol | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Todd Ruppar, PhD, RN, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No